CLINICAL TRIAL: NCT02994472
Title: Gastric Emptying: in Vivo Studies in Healthy Volunteers (Using Scrambled Egg and Porridge) to Determine Reliable Normal Ranges
Brief Title: Gastric Emptying: in Vivo Studies in Healthy Volunteers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sandwell & West Birmingham Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Shazmeen Hansrod, Clinical Scientist, Sandwell & West Birmingham Hospitals NHS Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 205705
Record Dates: First submitted 2016-12-08; First posted 2016-12-15 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Gastric Disease
MeSH Terms: conditions — Stomach Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy volunteers (Experimental): Each participant will have to eat scrambled egg on day 1 and porridge on day 2; both meals will contain the radioactive tracer 99mTc-DTPA.
  Participants will be scanned by a trained technologist. The scans will be carried out using a General Electric, Discovery 360 Gamma Camera.The scanning process will take approximately three hours in total, however the imaging will be carried out in stages.
  Interventions: Radiation: Gastric emptying scintigraphy using 99mTc-DTPA

INTERVENTIONS:
Radiation: Gastric emptying scintigraphy using 99mTc-DTPA

SUMMARY:
The Investigators institution has used a meal consisting of mashed potato, peas and Beanfeast (soya mince) for gastric emptying studies for a number of decades. Validation of the study method was purportedly performed when the study was first implemented at the hospital, however no historical data has been found. The current normal ranges are also unsubstantiated. There is scientific justification for this research because in vivo studies are instrumental to the validation of a new procedure. There is a need for a meal preparation that is palatable and meets dietary requirements (vegetarian, gluten free e.t.c.) of patients as the diagnosis depends on ingestion of the radiolabelled meal. In addition, reliable normal ranges will ensure that the clinical diagnosis is accurate. Scientific justification extends beyond the local department as publishing the data acquired will allow other hospitals to adopt the same test meals and normal ranges, leading to standardisation of the clinical protocol employed across the UK. Since the investigators institution are recognised as the leading Nuclear Medicine GI centre in the UK and have previously carried out audits and in vitro testing in the area of gastric emptying, it seems fit that they should lead the national change in protocol.

The proposed study will involve recruitment of healthy volunteers who will eat a meal containing 10MBq of a radioactive tracer. They will be subsequently scanned using a gamma camera with imaging lasting no more than 3 hours in total. Approximately 40 healthy volunteers (18-70 years old, no history of gastrointestinal problems or other serious health issues e.g. diabetes and pregnant women are excluded) will be recruited and the studies will be conducted on site i.e. within the Nuclear Medicine department at City hospital.

DETAILED DESCRIPTION:
After the ingestion and subsequent passage of solid or liquid material into the stomach, the gastric contents will undergo gastric emptying from the stomach into the intestine. The rate of gastric emptying can be very variable and will depend on the presence of gastric pathology or defect, composition and volume of the gastric contents and may even be influenced by factors such as gender and reproductive status. Gastric motility disorders such as gastroparesis and dumping syndrome can affect the rate of gastric emptying and thus warrant the quantitative assessment of emptying. Gastroparesis is a disorder of the stomach characterised by delayed gastric emptying in the absence of any mechanical obstruction and can be further categorised based on severity; mild gastroparesis (where symptoms can be easily controlled), compensated gastroparesis (partial control with use of medication and dietary adjustments) and gastric failure (symptoms are not controllable). Dumping syndrome occurs as a result of rapid gastric emptying which is usually associated with hypermotility of the stomach. It manifests as either early or late dumping syndrome, both of which have distinct physiological bases and clinical presentations.

Typical symptoms of delayed emptying include nausea, vomiting, abdominal pain and abdominal fullness after eating whilst diarrhoea, weakness and light headedness after meal times are common symptoms of rapid emptying. In the Nuclear Medicine department at City Hospital (Birmingham), patients referred for imaging are usually diabetics suffering from feelings of bloatedness after eating and occasional vomiting. Most patients studied are clinically diagnosed with gastroparesis associated with diabetes (where the vagus nerve responsible for controlling movement of food through the digestive tract stops functioning). Dumping is rarely reported as there is an effective tablet treatment for the disorder that usually eases the symptoms. (This includes octreotide therapies which can exert an effect through various mechanisms such as delaying transit, inhibiting the release of gut peptides and impaired fluid secretion). If left untreated gastroparesis can make diabetes worse by making it more difficult to manage blood glucose. Assessment of gastric emptying rate is therefore an important part of diagnosis.

Gastric emptying scintigraphy is a non-invasive diagnostic tool that is used in Nuclear Medicine to study the emptying of contents into the stomach. This form of scintigraphic examination is reproducible, simple to perform, accurate, quantitative and exposes the patient to only a very small radiation dose. It has been significantly optimised and refined over the years and is now well established as the standard method for evaluating gastric emptying. As the 'gold standard' gastric emptying scintigraphy is usually the first stage of the diagnostic journey for a patient, although some may have had a prior endoscopy (usually in cases of severe vomiting).

The procedure is known to vary between institutions, however will usually involve binding of a radiotracer to a solid or liquid meal which is then administered orally. This is followed by positioning of the patient in front of a camera and continuous or intermittent imaging is performed. Data is acquired over a length of time (usually 1-2 hours) and the data subsequently analysed to determine the half emptying time (i.e. the time required for the stomach to empty 50% of the ingested meal) which is then compared to established normal ranges (i.e. normal emptying rate expected for healthy individual). The current radioactive meal used for the study consisting of mashed potato, peas and Beanfeast (soya mince) is not particularly palatable, does not meet the dietary requirements of some patients (e.g. gluten/wheat free) and is difficult to prepare. In addition, in-house in vitro studies have found the current meal to be inferior to other meal preparations. Subjecting the radioactive meal to simulated conditions of the stomach has found that the radiolabel retention was significantly better in other meals such as scrambled egg and porridge.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female participants
* Age range of 18-70 years old
* All ethnicities/socio economic grouping
* Participants living outside local area (but within UK) included (but excessive travel may not be reimbursed)

Exclusion Criteria:

* Outside stated age range
* Outside the UK
* Have Diabetes or severe gastrointestinal symptoms such as vomiting or diarrhoea.
* Have a gastric motility disorder
* Pregnant women (If a participant becomes pregnant before their first test, they will be withdrawn from the study, If a participant becomes pregnant between the two tests, they will not be eligible for the second test but data collected from the first test may still be used for analysis).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Participants subject to Gastric Emptying Scintigraphy, emptying time expressed relative to normal range. | 1-2 years

CONTACTS AND LOCATIONS:
Overall Officials: Shazmeen Hansrod, Principal Investigator — Sandwell and West Birmingham Hospitals NHS Trust

IPD SHARING:
Plan to Share IPD: No
Individual Participant data will not be made available to other researchers.